CLINICAL TRIAL: NCT04502355
Title: Voriconazole-Induced QT Interval Prolongation: A Prospective Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Rabin Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 0483-16-RMC
Record Dates: First submitted 2020-08-04; First posted 2020-08-06 (Actual); Last update posted 2020-08-06 (Actual); Status verified 2020-08

CONDITIONS: Voriconazole Induced QT Interval Prolongation
Keywords: voriconazole, ECG, arrhythmia
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The antifungal voriconazole is effective for the treatment of invasive fungal infections in immunocompromised patients. A serious adverse reaction is QT interval prolongation, which may precede life-threatening arrhythmias, such as torsades de pointes. Although ventricular arrhythmias are mentioned as a possible adverse effect of voriconazole, thus far, the incidence and clear recommendations for QT follow-up have not been published. This prospective observational study aimed at describing the incidence of voriconazole induced- QT interval prolongation in the pediatric population and determine the risk factors for this phenomenon.

ELIGIBILITY:
Inclusion Criteria:

* oral or IV treatment with voriconazole

Exclusion Criteria:

* No data prior to initiation of voriconazole treatment on QT interval (baseline ECG)
* Renal insufficiency or dialysis treatment

Max Age: 20 Years | Sex: All
Age Groups: Child, Adult
Study Population: Children aged 0-20 years treated with oral or IV voriconazole at the Schneider Children's Medical Center from Oct 31st 2016.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2016-10-31 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
QT interval prolongation | up to three months of treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Schneider childrens medical center of Isreal, Petah Tikva, Israel

IPD SHARING:
Plan to Share IPD: Undecided